CLINICAL TRIAL: NCT05492149
Title: Pulmonary Rehabilitation for COPD Patients: Can Performance Predict Exacerbation?
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00210-43
Record Dates: First submitted 2022-07-26; First posted 2022-08-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD; COPD Exacerbation; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary rehabilitation group: Patients referred for a pulmonary rehabilitation program will be follow up.
  Interventions: Other: Performance follow-up

INTERVENTIONS:
Other: Performance follow-up — Diary performance during rehabilitation will be collected and a CAT questionnaire will be completed by the patient.

SUMMARY:
The aim of pulmonary rehabilitation is to improve exercise capacity and reduce dyspnoea. As well as improving the patient's overall condition, pulmonary rehabilitation provides a means to monitor the patient regularly. During physical exercise, the increased activity of the muscle system increases cardiac and respiratory output. If the patient's respiratory status deteriorates, as occurs, for example, before the onset of an exacerbation, exercise capacity could be reasonably expected to reduce. The investigators hypothesised, therefore, that changes in the physical capacity of patients with COPD during a rehabilitation session could provide a predictive indication regarding the risk of occurrence of exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* COPD patients

Exclusion Criteria:

* Patients who not performed not at least 5 sessions of the pulmonary rehabilitation program
* Occurence of an adverse event that prevents further rehabilitation
* Exacerbation in the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients who referred to a pulmonary rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the decrease of performance during pulmonary rehabilitation session and the occurrence of pulmonary exacerbation. | From admission to the program or first documented session ; to completion of the pulmonary rehabilitation program or occurrence of an exacerbation, up to 104 weeks.
  The change in performance rehabilitation of patients between the last session will be screen when a patients will be admitted to hospital for a COPD exacerbation.

SECONDARY OUTCOMES:
Correlation between the decrease of performance during pulmonary rehabilitation session and the COPD Assessment Test (CAT) questionnaire score. | Through study completion, at every pulmonary rehabilitation session ; to completion of the pulmonary rehabilitation program or occurrence of an exacerbation, up to 104 weeks.
  The change in performance rehabilitation of patients between the last session will be screen and compared to a COPD Assessment Test (CAT) questionnaire score.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Montivilliers, Groupe Hospitalier Du Havre, France

IPD SHARING:
Plan to Share IPD: Undecided
by contact the correspondent author